CLINICAL TRIAL: NCT06036095
Title: Optimizing Anesthesia to Prevent Postoperative Cognitive and Functional Decline in Older Adults: A Randomized Controlled Trial
Brief Title: Total Intravenous Versus Inhalational Anesthesia- A Geriatric Anesthesia Study
Acronym: TIVA GAS
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Katie J. Schenning, Associate Professor, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: STUDY00024667
Record Dates: First submitted 2023-04-18; First posted 2023-09-13 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: Neurocognitive Disorders; Anesthesia; Post-operative Delirium; Post-operative Cognitive Dysfunction
MeSH Terms: conditions — Neurocognitive Disorders; Emergence Delirium | interventions — Sevoflurane; Propofol; Anesthesia, Intravenous

STUDY DESIGN:
Intervention Model Description: This single-center, 1:1 randomized, double-blind (patient & outcome assessor) clinical trial will compare inhalational (sevoflurane) vs. intravenous (propofol) anesthesia on POD, POCD, functional status, PROs, and biomarkers in patients ≥ 70 years undergoing elective, inpatient, non-cardiac surgery at Oregon Health & Science University.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Inhalational Anesthesia (Active Comparator): Inhalational maintenance of anesthesia group using sevoflurane
  Interventions: Drug: Sevoflurane
- Intravenous Anesthesia (Active Comparator): Intravenous maintenance of anesthesia group using propofol
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Sevoflurane — Inhalational maintenance of anesthesia group using sevoflurane
  Other Names: Inhalational Anesthesia
  Arms: Inhalational Anesthesia
Drug: Propofol — Intravenous maintenance of anesthesia group using propofol
  Other Names: Intravenous Anesthesia
  Arms: Intravenous Anesthesia

SUMMARY:
Traditionally, general anesthesia is maintained with inhalational anesthesia (GAS), but there is a gap in knowledge regarding whether intravenous anesthesia (IV) can prevent deleterious postoperative outcomes in the geriatric surgical population. The goal of this clinical trial is to determine whether intravenous anesthesia (IV) leads to a decreased incidence of postoperative delirium (POD), postoperative cognitive dysfunction (POCD), and functional decline, and improved patient-reported outcomes (PROs) in older adults undergoing non-cardiac surgery when compared to the standard inhalational anesthesia (GAS). This single-center, 1:1 randomized, double-blind (patient & outcome assessor) clinical trial will compare inhalational vs. intravenous anesthesia on POD, POCD, functional status, patient-reported outcomes (PROs), and blood-based biomarkers in older patients undergoing elective, inpatient, non-cardiac surgery. Upon enrollment, 260 women and men ≥ 70 years undergoing elective noncardiac surgery under general anesthesia will be randomized to 2 groups: TIVA or GAS.

DETAILED DESCRIPTION:
Aim 1: Determine the effects of intravenous vs. inhalational anesthesia on incidence of postoperative delirium and postoperative cognitive dysfunction in older adults undergoing non-cardiac surgery.

Hypothesis: Intravenous anesthesia is associated with a lower incidence of POD and POCD compared to inhalational anesthesia.

Primary outcomes: Incidence of postoperative delirium and postoperative cognitive dysfunction Secondary outcomes: delirium severity, delirium duration Aim 2: Determine the effects of intravenous vs. inhalational anesthesia on incidence of postoperative functional decline and patient-reported outcomes in older adults undergoing non-cardiac surgery.

Hypothesis: Intravenous anesthesia is associated with a lower incidence of postoperative functional decline and improved patient-reported outcomes (PROs) compared to inhalational anesthesia.

Primary outcomes: Incidence of postoperative functional decline; patient-reported outcome scores Aim 3: Determine the effects of intravenous vs. inhalational anesthesia on blood phosphorylated tau 181 (p-tau181) and other blood biomarkers in older adults undergoing non-cardiac surgery.

Hypothesis 1: Elevated preop blood p-tau181 is associated with increased POD and POCD; Hypothesis 2: Postoperative increase in blood p-tau181 is greater with GAS relative to IV; Hypothesis 3: Postop increases in blood biomarkers of neuroinflammation and AD pathology are greater with GAS relative to IV.

Primary outcomes: preoperative levels of blood p-tau181 and change in levels from preoperative baseline to postoperative.

Secondary outcomes: Other candidate biomarkers include those previously implicated in POD or POCD: p-tau217, Aβ,54 NF-L,55 High mobility group box protein 1 (HMGB1),60 S100β,76 interleukin (IL)-6,58 IL-1β,22 IL-10,46 tumor necrosis factor (TNF)-α,22 CCL2,62 and glial fibrillary acidic protein (GFAP).77

ELIGIBILITY:
Inclusion criteria:

* Men and women ≥ 70 years
* Sufficient vision and hearing to complete all tests
* Proficient in spoken and written English
* Scheduled for elective, inpatient, noncardiac surgery, expected to last at least 120 minutes requiring general anesthesia

Exclusion criteria:

* Urgent or emergent surgery
* Diagnosed dementia (or MoCA<19)
* History of Parkinson's disease, major psychiatric disease (Schizophrenia), or severe traumatic brain injury
* Ongoing alcohol or substance abuse (per DSM V criteria)
* Allergy to propofol or sevoflurane
* Personal or family history of malignant hyperthermia
* Planned postoperative intubation
* Brain surgery
* Surgery requiring TIVA or GAS (i.e. cases involving neuromonitoring)
* Surgical procedure requiring general anesthetic occurring within 3 months (before or after) surgical date
* Any patient or perioperative factor considered a contraindication to randomization to either experimental group by the surgeon or anesthesiologist.

Ages: 70 Years to 110 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2023-08-14 (Actual); Primary Completion 2027-03-15 (Estimated); Study Completion 2027-03-15 (Estimated)

PRIMARY OUTCOMES:
Effects of intravenous vs. inhalational anesthesia on incidence of postoperative delirium in older surgical patients with the 3D-Confusion Assessment Method (3D-CAM-S) and the CAM-ICU-7. | through postoperative day 3
  Incidence of postoperative delirium with the 3D-Confusion Assessment Method (3D-CAM) in non-intubated patients and the CAM-ICU-7 in intubated patients. Delirium will be assessed postoperative in PACU and twice daily on postoperative days 1-3 while the patient is in the hospital.
Determine the effects of intravenous vs. inhalational anesthesia on the incidence of postoperative neurocognitive disorder in older adults undergoing non-cardiac surgery using neuropsychiatric composite score. | Change from preoperative baseline to one year.
  Postoperative neurocognitive disorder. Change from preoperative baseline cognitive dysfunction using neuropsychiatric composite score. Battery of neuropsychological tests: Animal Verbal Fluency Test, Trail Making Test A & B, Digit Symbol Test, Logical Memory Immediate & Delayed Recall, and CERAD Word List Immediate and Delayed recall. MASQ will be used for subjective cognitive decline. Functional status will be measured by FAQ.

SECONDARY OUTCOMES:
Determine the effects of intravenous vs. inhalational anesthesia on incidence of delirium duration (days) and severity, measured by 3D-CAM-S, and CAM-ICU-7 in older adults undergoing non-cardiac surgery. | through postoperative day 3
  delirium severity and duration. Delirium will be assessed postoperative in PACU and twice daily on postoperative days 1-3.
Effects of intravenous vs. inhalational anesthesia on levels of blood phosphorylated tau 181 (p-tau181) in older surgical patients.. Change from preoperative baseline blood p-tau181 to postoperative day 1, 3 months and 12 months. | Change from baseline through one year.
  change in levels of preoperative levels of blood p-tau181 from preoperative baseline to 12 months postoperative
Determine the effects of intravenous vs. inhalational anesthesia on incidence of postoperative functional decline using ADL, FAQ, and FRAIL in older adults undergoing non-cardiac surgery. | Change from baseline through one year
  Incidence of postoperative functional decline. Change from preoperative baseline postoperative functional decline to postoperative 12 months.
Determine the effects of intravenous vs. inhalational anesthesia on patient-reported outcomes (PROMIS-29+2 Profile v2.1) in older adults undergoing non-cardiac surgery. | Change from baseline through one year
  patient-reported outcome scores, PROMIS-29+2 Profile v2.1 (PROPr) assesses patient-reported measures of anxiety, depression, fatigue, pain interference, physical function, sleep disturbance, participation in social activities, pain, and cognition. Measured at preoperative baseline, 3 months postoperatively, and 12 months postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Katie J. Schenning, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: Yes
In order to promote advancement of this field of study, we will make data generated from this project available. Participants will sign a data repository consent form so de-identified data is able to be maintained indefinitely on secure servers at Oregon Health & Science University. This will enable us to combine these data with other datasets for future analyses, and to share with collaborators and other interested scientists. Other researchers would sign a data use agreement and then receive the de-identified data requested.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code